CLINICAL TRIAL: NCT02941198
Title: Comparative of Two Devices (Conventional Intrauterine Devices (Cu T380 A)/Frameless Intrauterine Devices (GyneFix)) for Postpartum Immediate Contraception in Cesarean Deliveries
Brief Title: Postpartum Immediate Contraception in Cesarean Deliveries-Comparison of Two Intrauterine Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Ahmet Eser, medical doctor, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 110
Record Dates: First submitted 2016-10-12; First posted 2016-10-21 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-01

CONDITIONS: Intrauterine Systems; Postpartum Immediate Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gynefix (Active Comparator): The GyneFix® 200 IUD(frameless iud) is only 2 cm long. Its small surface area is 1/3 of that of the conventional T-shaped IUDs such as TCu380A
  Interventions: Device: GyneFix
- Cu T380a (Active Comparator): conventional T-shaped IUDs (TCu380A)which has a frame will be placed into the uterus after placental extraction
  Interventions: Device: Cu T380 A

INTERVENTIONS:
Device: GyneFix — The fiber is fixed to the anchoring thread by means of a stainless steel clip 1 cm from the upper part of the anchoring knot. The anchoring knot is implanted into the myometrium of the uterus thus permanently securing the implant in the uterine cavity
  Other Names: Gynefix(frameless intrauterine devices)
  Arms: Gynefix
Device: Cu T380 A — Cu T380 A will be inserted into the uterus
  Other Names: Copper T 380a
  Arms: Cu T380a

SUMMARY:
To compare two intrauterine systems in order to avoid complications originating from short pregnancy interval and undesired pregnancies in the early postpartum period.

DETAILED DESCRIPTION:
The patients admitting to Zeynep Kamil Research and Training Hospital for caesarean delivery will be included in the study. There will be two computer based randomized groups. The investigators expect that both groups will have 100 cases. First group will be treated with conventional intrauterine devices (Cu T380 A) while the second group will be treated with frameless intrauterine devices (GyneFix). The participants will be informed about postpartum unplanned pregnancies and the complications of short pregnancy interval. Participants will also be informed about possible complications of having an intrauterine device and that there may be a possibility of failure.The participants who choose to participate in the study will be divided into two groups by computer based randomization and one of the systems will be applied. After the participants read and sign the informed consent form, the intrauterine device will be applied postplacental up to 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* The patients who read and sign the informed consent form.

Exclusion Criteria:

* The patient who has more than 6 cm dilatation, prolonged premature rupture of the membranes (more than 12 hours), chorioamnionitis, and kongenital or acquired haemorragic diathesis will be excluded from the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
expulsion rates | The patients will be seen postoperative 6th week
  expulsion is the major obstacle for intrauterin devices when using immediate postpartum.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by conventional intrauterine devices (Cu T380 A) and frameless intrauterine devices (GyneFix) | The patients will be seen postoperative 6th week
  there are some effects due to intrauterin devices. we want to compare the differences between two devices

CONTACTS AND LOCATIONS:
Overall Officials: ceren ünal, m.d., Principal Investigator — medical doctor
Locations (1):
- Zeynep Kamil Maternity and Children's Training and Research Hospital, Department of Obstetrics and Gynecology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hooda R, Mann S, Nanda S, Gupta A, More H, Bhutani J. Immediate Postpartum Intrauterine Contraceptive Device Insertions in Caesarean and Vaginal Deliveries: A Comparative Study of Follow-Up Outcomes. Int J Reprod Med. 2016;2016:7695847. doi: 10.1155/2016/7695847. Epub 2016 Aug 17. PMID 27631023
- [Background] Lopez LM, Bernholc A, Hubacher D, Stuart G, Van Vliet HA. Immediate postpartum insertion of intrauterine device for contraception. Cochrane Database Syst Rev. 2015 Jun 26;2015(6):CD003036. doi: 10.1002/14651858.CD003036.pub3. PMID 26115018
- [Background] Singal S, Bharti R, Dewan R, Divya, Dabral A, Batra A, Sharma M, Mittal P. Clinical Outcome of Postplacental Copper T 380A Insertion in Women Delivering by Caesarean Section. J Clin Diagn Res. 2014 Sep;8(9):OC01-4. doi: 10.7860/JCDR/2014/10274.4786. Epub 2014 Sep 20. PMID 25386484
- [Background] Bhutta SZ, Butt IJ, Bano K. Insertion of intrauterine contraceptive device at caesarean section. J Coll Physicians Surg Pak. 2011 Sep;21(9):527-30. PMID 21914407